CLINICAL TRIAL: NCT06083246
Title: Efficacy of Hybenix and Chlosite Gels in Peri-implantitis Sites: a 9-month Randomized Clinical Trial.
Brief Title: Clinical Efficacy of Hybenix vs Chlosite Gels in Peri-implantitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-IMPLGEL
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Peri-Implantitis
Keywords: Chlorhexidine; Hybenix gel; Domiciliary treatments
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybenix gel (Experimental): Clinical application of Hybenix gel.
  Interventions: Other: Hybenix gel
- Chlosite (Active Comparator): Clinical application of Chlosite gel.
  Interventions: Other: Chlosite gel

INTERVENTIONS:
Other: Hybenix gel — Clinical application of Hybenix gel after professional dental hygiene of peri-implant mucositis sites.
  Arms: Hybenix gel
Other: Chlosite gel — Clinical application of Chlosite gel after professional dental hygiene of peri-implant mucositis sites.
  Arms: Chlosite

SUMMARY:
The present study is a randomized clinical trial (RCT). Patients responding to the inclusion criteria will be included. The following peri-implant indexes will be collected: Bleeding On Probing, Gingival Bleeding Index, Marginal Mucosal Conditions (swelling and erythema), Suppuration, Mucosal margin migration, PPD Probing Pocket Depth, Plaque Index, Bleeding Score, radiographic bone loss.

After the peri-implant evaluation, patients will undergo supragingival and subgingival professional oral hygiene of both arches performed with ultrasonic instrumentation with PEEK inserts, manual instrumentation with teflon curettes and air polishing with glycine powder.

After that, the sample will be randomly divided into 2 groups based on thein-office assigned treatment:

* Chlosite® gel application in the peri-implant sulcus
* Hybenix® gel application for 30 s followed by rinsing of the peri-implant sulcus.

The study will last 9 months. Patients will be visited at: T0, after 1 month from T0 (T1), after 3 months (T2), after 6 months (T3) and after 9 months (T4).

In each time frame, indexes collection and nonsurgical debridement will be performed.

DETAILED DESCRIPTION:
The present study is designed as a randomized clinical trial (RCT) to evaluate the clinical efficacy of two adjuvant gels in the treatment of perimplantitis.

Patients responding to the inclusion criteria will be included in the study. The following peri-implant indexes will be collected:

* BOP (Bleeding On Probing)
* GBI (Gingival Bleeding Index)
* Marginal Mucosal Conditions (swelling and erythema)
* Suppuration
* Mucosal margin migration
* PPD (Probing Pocket Depth)
* PI (Plaque Index)
* BS (Bleeding Score)
* Radiographic bone loss

After the peri-implant evaluation, patients will undergo supragingival and subgingival professional oral hygiene of both arches performed with ultrasonic instrumentation with PEEK inserts, manual instrumentation with teflon curettes and air polishing with glycine powder.

After that, the sample will be randomly divided into 2 groups based on thein-office assigned treatment:

* Chlosite® gel application in the peri-implant sulcus
* Hybenix® gel application for 30 s followed by rinsing of the peri-implant sulcus.

The study will last 9 months. Patients will be visited at: T0, after 1 month from T0 (T1), after 3 months (T2), after 6 months (T3) and after 9 months (T4).

In each time frame, indexes collection and nonsurgical debridement will be performed.

ELIGIBILITY:
Inclusion Criteria:

- Presence of at least one peri-implant site with perimplantitis diagnosed according to the latest Classification of Periodontal and Peri-Implant Diseases and Conditions [Berglundh et al., 2018]

Exclusion Criteria:

* Patient with cardiac pacemaker
* Patients suffering from psychological, neurological or psychiatric disorders
* Patients suffering from systemic, metabolic or autoimmune diseases
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Change in BOP - Bleeding On Probing | Baseline, 1, 3, 6 and 9 months.
  Dichotomous scoring (yes/no)
Change in GBI - Gingival Bleeding Index (percentage) | Baseline, 1, 3, 6 and 9 months.
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 6 sites.
  The number of bleeding sites is divided per the total number of probed sites; the ratio is multiplied X 100.
Change in marginal mucosa condition | Baseline, 1, 3, 6 and 9 months.
  Scoring criteria:
  0: normal mucosa
  1. minimal inflammation with color change and minor edema
  2. moderate inflammation with redness, edema and glazing
  3. severe inflammation with redness, edema, ulceration and spontaneous bleeding without probing
Change in suppuration | Baseline, 1, 3, 6 and 9 months.
  Dichotomous scoring (yes/no)
Marginal mucosal migration | Baseline, 1, 3, 6 and 9 months.
  Dichotomous scoring (yes/no)
Probing Depth | Baseline, 1, 3, 6 and 9 months.
  Evaluation (in mm) of the depth of the mucosal sulcus, through a millimeter periodontal probe; it is detected from the mucosal margin to the bottom of the peri-implant sulcus, evaluated at 6 sites.
Change in BS - Bleeding Score | Baseline, 1, 3, 6 and 9 months.
  Scoring criteria:
  0: no bleeding
  1. isolated visible spots
  2. blood forms a confluent red line on mucosal margin
  3. heavy or profuse bleeding
Change in PI - Plaque Index (percentage) | Baseline, 1, 3, 6 and 9 months.
  Evaluation of the presence of plaque on the 4 surfaces of teeth on the total amount of dental surfaces.
Change in Radiographic bone loss (percentage) | Baseline, 1, 3, 6 and 9 months.
  Quantitative evaluation of the bone loss evaluated on intraoral x-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MSc, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.